CLINICAL TRIAL: NCT02185508
Title: Intra-operatory Neurophysiological Monitoring Changes as a Predictive Clinical Outcome Measure in Radiculopathy Associated to Lumbar Disk Disease. Two Years Follow-up
Brief Title: Intra-operatory Neurophysiological Monitoring Changes as a Predictive Clinical Outcome Measure in Lumbar Radiculopathy.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: American British Cowdray Medical Center (Other)
Responsible Party: Principal Investigator, Galvan Ernesto Eduardo, MD, American British Cowdray Medical Center
Other Study IDs: ABC-14-06
Record Dates: First submitted 2014-07-04; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Lumbar Disc Disease
Keywords: IONM; Lumbar Disk Disease; Degenerative Spine Disease; Radiculopathy; Intraoperative Neurophysiological Monitoring; Somatosensory Evoked Potentials; Electromyography
MeSH Terms: conditions — Intervertebral disc disease; Radiculopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Lumbar spine surgery with IONM: Patients diagnosed with 1 or 2 level lumbar disk disease and radicular symptoms who underwent decompressive surgery, and for whom IONM records exist.

SUMMARY:
The purpose of this study is to determine the relation among: (1) changes in voltage and amplitude of trans-operatory records obtained through the use of Intra-operative Neurophysiological Monitoring (IONM), and (2) clinical outcomes; of patients who underwent 1 or 2 levels surgical decompression at lumbar spine.

IONM is the use of real time neurophysiological techniques during spinal surgeries. The modalities included in this study are:

* Somatosensory evoked potentials (SSEPs).
* Trans-cranial electric motor evoked potentials (tceMEPs).
* Spontaneous electromyography (EMG).

Clinical outcome of the patients will be assessed through a careful evaluation of clinical data, as well as the application of three outcome scales:

* Oswestry Disability Index 2.1a
* Visual Analogue Scale for Pain
* Patient's Overall Impression of Change

DETAILED DESCRIPTION:
Radiculopathy associated to lumbar disk disease is one of the most common reasons for a spine surgeon to be consulted. The pathophysiology of degenerative spine disease is acknowledged as complex, involving a wide array of risk factors ranging from genetic polymorphisms, to behavioural characteristics. While conflicting opinions exist with regard the direction of treatment for lumbar disk disease, de-compressive surgery is currently the gold standard for patients in which protocols of physiotherapy and analgesics have failed to comply.

Intraoperative neurophysiological monitoring (IONM) is widely used in the practice of spine surgery as a mean of preventing and reducing severe complications inherent to surgical techniques like paraparesis, paraplegia and quadriplegia. Indeed, a great deal of funding and work have been devoted to research projects seeking to determine the impact of IONM in reducing these risks. The results of such projects have been notoriously interesting, and frequently opposing to each other. This has lead to an open debate on weather the use of IONM may or not be justified by better outcomes in patients who undergo such procedure. To our knowledge there is no study in the literature that has addressed the potential role of the IOM to predict the long-term outcome of the patient in therms of radicular symptoms improvement.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Lumbar Disk Disease
* Clinical Signs of Radiculopathy
* Undergoing neurological surgery of the spine

Exclusion Criteria:

* Previous neurological surgery of the lumbar spine
* More than 2 levels intervened at the surgery
* Serious post-operatory complications

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with lumbar disk disease with radiculopathy, undergoing neurological surgery of the spine at the ABC Neurological Center
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Electrophysiological changes measured through intraoperative neurophysiological monitoring. | Trans-operative
  Standard register electrodes where placed from L1 to L5 myotomes and dermatomes. Through trans-operative real time modalities (trans-cranial electric motor evoked potentials, somatosensory evoked potentials, and spontaneous electromyography) measurements on amplitude and voltage were recorded at the beginning and at the end of the spinal decompression. This change will be studied to determine its predictive power in the clinical long-term outcome of the patients.

SECONDARY OUTCOMES:
Visual analogue scale for pain | In the pre-operatory consult with the surgeon, and in the follow-up visits up to two years after the completion of the neurological surgery; the patient will be asked to complete the Visual Analogue Scale for Pain
  The visual analogue scale is a written survey used to assess the pain a person endures. The patient will select a number from one to ten to express the relative amount of pain she is suffering. Data collected throughout the study will be used as a clinical follow-up measure to be compared with that obtained through intraoperative neurophysiological monitoring. Approximate time of completion is <5 minutes; and no physical examination, nor additional pain may be experienced by completing such survey
Oswestry Disability Index 2.1a | In the pre-operatory consult with the surgeon, and in the follow-up visits up to two years after the completion of the neurological surgery; the patient will be asked to complete the Oswestry Disability Index 2.1a
  The Oswestry Disability Index 2.1a is a written survey used to quantify the amount of disability a person endures due to low-back pain. The patient will answer a series of 10 questions enquiring about experiences of her life, and how the pain she suffers affects the quality of these experiences. Data collected throughout the study will be used as a clinical follow-up measure to be compared with that obtained through intraoperative neurophysiological monitoring. Approximate time of completion is <5 minutes; and no physical examination, nor additional pain may be experienced by completing such survey.
Patient's Global Impression of Change Survey | In the follow-up visits up to two years after the completion of the neurological surgery, the patient will be asked to complete the Patient's Global Impression of Change Survey
  The Patient's Global Impression of Change Survey is a written survey used to quantify the amount of improvement a person perceives for herself after receiving a certain treatment. The patient will select from a list of previously defined statements, the one that best describes her impression of change after the surgery, and will select a number ranging from one to ten representing her perception of improvement. Data collected throughout the study will be used as a clinical follow-up measure to be compared with that obtained through intraoperative neurophysiological monitoring. Approximate time of completion is <5 minutes; and no physical examination, nor additional pain may be experienced by completing such survey.

OTHER OUTCOMES:
General demographic, personal and biometrical data | In the pre-operatory consult with the surgeon, the patient will be asked to complete a survey enquiring about general demographic, personal and biometrical data
  The survey used to capture general demographic, personal and biometrical data is designed according to the stipulations of the Official Mexican Norm for the Clinical Record (NOM-004-SSA3-2012). The data obtained through such survey will help the surgeon in assessing the case of the patient. Some or all of this data may be used for analysis in this study, to be compared with the rest of the outcome measures. A privacy policy statement may be provided to the patient according to the Federal Law for the Protection of Personal Data in Possession of Particulars (Ley Federal de Protección de Datos Personales en Posesión de los Particulares). Regardless of such formality, the privacy of the patient will be assured throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto De Leo Vargas, MD, Study Director — American British Cowdray Medical Center; Maximino Tellez, MD, Study Chair — American British Cowdray Medical Center; Ildefonso Muñoz Romero, MD, Study Chair — American British Cowdray Medical Center; Miguel Angel Collado Corona, MD, Study Chair — American British Cowdray Medical Center; Leopoldo Torres Vyera, MD, Study Chair — American British Cowdray Medical Center; Christian Cerecedo, MD, Study Chair — American British Cowdray Medical Center; Eduardo Galvan Hernandez, MD, Principal Investigator — American British Cowdray Medical Center
Locations (1):
- American British Cowdray Medical Center, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Koerner JD, Glaser J, Radcliff K. Which Variables Are Associated With Patient-reported Outcomes After Discectomy? Review of SPORT Disc Herniation Studies. Clin Orthop Relat Res. 2015 Jun;473(6):2000-6. doi: 10.1007/s11999-014-3671-1. PMID 24818737
- [Background] Sabnis AB, Diwan AD. The timing of surgery in lumbar disc prolapse: A systematic review. Indian J Orthop. 2014 Mar;48(2):127-35. doi: 10.4103/0019-5413.128740. PMID 24741132
- See also: Para mas informacion sobre hernias de disco, porfavor visite la siguiente pagina de internet: — http://www.nlm.nih.gov/medlineplus/spanish/ency/article/000442.htm
- See also: For more information on disk hernias, please visit the following web page: — http://www.nlm.nih.gov/medlineplus/ency/article/000442.htm